CLINICAL TRIAL: NCT00239655
Title: A Randomized, Double-Blind Placebo Controlled, Parallel Groups Study to Assess the Effects of MK0812 on Disease Activity in Patients With Relapsing-Remitting Multiple Sclerosis as Measured by MRI
Brief Title: A Study to Assess the Effects of MK0812 on Disease Activity in Patients With Relapsing-Remitting Multiple Sclerosis as Measured by Magnetic Resonance Imaging (MRI)(0812-003)(COMPLETED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0812-003; MK0812-003; 2005_087
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0812

SUMMARY:
The purpose of this study is to test MK0812 on disease activity in patients with relapsing-remitting MS. Disease modifying activity will be assessed by measurement of brain lesions via MRI brain scans and an open label extension is offered.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically definite relapsing-remitting MS onset within last 10 years and have had at least 1 objective clinical exacerbation in the last year OR a recent clinically isolated syndrome suggestive of MS occurring 3-12 months before screening
* Patients must be relatively healthy

Exclusion Criteria:

* Patient has primary progressive MS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2004-08; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Accrual rate of new GD-enhancing lesions as assessed by MRI | 3 Months

SECONDARY OUTCOMES:
Volume and cumulative number of new persistent Gd-enhancing lesions | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC